CLINICAL TRIAL: NCT01200914
Title: Placement of Covered Stents to Treat Hemodialysis Access Stenosis in the Cephalic Arch and Central Veins
Brief Title: Covered Stents to Treat Hemodialysis Access Stenoses in the Cephalic Arch and Central Veins
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor recruitment
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Dheeraj Rajan, Head and Associate Professor, Division of Vascular & Interventional Radiology, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORE-001
Record Dates: First submitted 2010-09-10; First posted 2010-09-14 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Renal Failure
Keywords: Hemodialysis; Fistula; Angiograph; Angiogram
MeSH Terms: conditions — Renal Insufficiency; Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 'PTA without use of the GORE VIABAHN' (Active Comparator): Subjects randomized to 'PTA alone without use of the GORE VIABAHN' will receive the standard of care treatment which is Percutaneous Transluminal Angioplasty without the use of the 'GORE VIABAHN® Endoprosthesis with Heparin Bioactive Surface'
  Interventions: Procedure: PTA alone without use of the GORE VIABAHN
- PTA with covered stent (Experimental): Subjects randomized to PTA with covered stent will receive Percutaneous Transluminal Angioplasty followed by the delivery of a 'GORE VIABAHN® Endoprosthesis with Heparin Bioactive Surface' .
  Interventions: Device: GORE VIABAHN® Endoprosthesis with Heparin Bioactive Surface

INTERVENTIONS:
Device: GORE VIABAHN® Endoprosthesis with Heparin Bioactive Surface — The 'GORE VIABAHN® Endoprosthesis with Heparin Bioactive Surface' will be deployed at the brachiocephalic stenosis.
  Other Names: Covered stent
  Arms: PTA with covered stent
Procedure: PTA alone without use of the GORE VIABAHN — Subject will receive standard of care PTA alone at the brachiocephalic stenosis without deployment of the'GORE VIABAHN® Endoprosthesis with Heparin Bioactive Surface'
  Arms: 'PTA without use of the GORE VIABAHN'

SUMMARY:
Balloon angioplasty is used to open up a narrowing that forms in hemodialysis fistula. Two areas of particular problems are the terminal portion of the cephalic vein near the shoulder and the central veins in the chest. Although angioplasty is standard of care the treated narrowed segments of vein mostly renarrow within 3 months requiring retreatment to keep your dialysis access functional. Recently there has been introduction of a new technology called a covered stent graft. Initial studies suggest that placing this device across the area of narrowing leads to dialysis access staying open longer and needing less angioplasty treatments.

This study is designed to compare angioplasty (standard of care) versus using a covered stent graft. The investigators will then look at the dialysis records and future fistulograms to see if there is decreased flow through the fistula at 3, 6 and 12 months after the initial procedure.

DETAILED DESCRIPTION:
This is a randomized, prospective, unblinded study with 1:1 randomization. Both groups will undergo PTA of stenotic lesion and patients will be randomized such that 50% will receive a covered stent in addition to the PTA. Patients will be followed at 3, 6, and 12 months post-procedure. Follow-up will be conducted with either angiographic and/or transonic measurements.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patient with a mature forearm or upper arm access that was created > 2 months before enrollment in study.
* The patient is ≥ 18 years of age.
* The patient has a reasonable expectation of remaining on hemodialysis for 12 months.
* The patient or his/her legal guardian understands the study and is willing and able to comply with follow-up requirements.
* The patient or his/her legal guardian is willing to provide informed consent.
* The patient has lesions that meet the angiographic inclusion / exclusion criteria and induce clinical, hemodynamic or functional abnormality.

Exclusion Criteria:

* The patient has a known or suspected systemic infection.
* The patient has a known or suspected infection of the hemodialysis access and / or bacteremia.
* The patient is currently taking maintenance immunosuppressant medication such as rapamycin, mycophenolate or mycophenolic acid, prednisone (>10 mg per day), cyclosporine, tacrolimus, or cyclophosphamide.
* The patient has known bleeding disorder (e.g., hemophilia or von Willebrand's disease).
* The patient has known sensitivity to heparin.
* The patient is scheduled for a live donor kidney transplant.
* The patient is enrolled in another investigational study or another access maintenance trial
* The patient has comorbid conditions that may limit their ability to comply with the follow-up requirements.
* Life expectancy is ≤ 24 months.
* The patient has an untreatable allergy to radiographic contrast material.
* The patient is pregnant.
* In the opinion of the operating physician, the patient's hemodialysis access circuit is unsuitable for endovascular treatment.
* The patient's access is planned to be abandoned within 1 year.
* The patient has indwelling catheters (dialysis, pacemakers, ports).
* The patient has a central vein stent that would lead to jailing of the internal jugular vein.
* The patient experiences angioplasty-induced venous rupture.
* The patient has a flow limiting dissection after angioplasty.
* The patient's hemodialysis access is thrombosed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Target lesion primary patency at 3, 6, and 12 months | 1 year

SECONDARY OUTCOMES:
Target lesion secondary patency at 3, 6, and 12 months, access circuit primary and secondary patency at 3, 6, and 12 months, anatomic, clinical, and procedural success. Adverse events through 1 month | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dheeraj Rajan, M.D., Principal Investigator — Physician
Locations (1):
- Universtiy Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Gray RJ, Sacks D, Martin LG, Trerotola SO; Society of Interventional Radiology Technology Assessment Committee. Reporting standards for percutaneous interventions in dialysis access. J Vasc Interv Radiol. 2003 Sep;14(9 Pt 2):S433-42. doi: 10.1097/01.rvi.0000094618.61428.58. No abstract available. PMID 14514859
- [Background] Sidawy AN, Gray R, Besarab A, Henry M, Ascher E, Silva M Jr, Miller A, Scher L, Trerotola S, Gregory RT, Rutherford RB, Kent KC. Recommended standards for reports dealing with arteriovenous hemodialysis accesses. J Vasc Surg. 2002 Mar;35(3):603-10. doi: 10.1067/mva.2002.122025. PMID 11877717
- [Background] Chang CJ, Ko PJ, Hsu LA, Ko YS, Ko YL, Chen CF, Huang CC, Hsu TS, Lee YS, Pang JH. Highly increased cell proliferation activity in the restenotic hemodialysis vascular access after percutaneous transluminal angioplasty: implication in prevention of restenosis. Am J Kidney Dis. 2004 Jan;43(1):74-84. doi: 10.1053/j.ajkd.2003.09.015. PMID 14712430
- [Background] Patel RI, Peck SH, Cooper SG, Epstein DM, Sofocleous CT, Schur I, Falk A. Patency of Wallstents placed across the venous anastomosis of hemodialysis grafts after percutaneous recanalization. Radiology. 1998 Nov;209(2):365-70. doi: 10.1148/radiology.209.2.9807560.
- [Background] Rajan DK, Clark TW. Patency of Wallstents placed at the venous anastomosis of dialysis grafts for salvage of angioplasty-induced rupture. Cardiovasc Intervent Radiol. 2003 May-Jun;26(3):242-5. doi: 10.1007/s00270-003-2706-x. PMID 14562971
- [Background] Haage P, Vorwerk D, Piroth W, Schuermann K, Guenther RW. Treatment of hemodialysis-related central venous stenosis or occlusion: results of primary Wallstent placement and follow-up in 50 patients. Radiology. 1999 Jul;212(1):175-80. doi: 10.1148/radiology.212.1.r99jl21175. PMID 10405739
- [Background] Vogel PM, Parise C. SMART stent for salvage of hemodialysis access grafts. J Vasc Interv Radiol. 2004 Oct;15(10):1051-60. doi: 10.1097/01.RVI.0000129915.48500.DC. PMID 15466790
- [Background] Rajan DK, Saluja JS. Use of nitinol stents following recanalization of central venous occlusions in hemodialysis patients. Cardiovasc Intervent Radiol. 2007 Jul-Aug;30(4):662-7. doi: 10.1007/s00270-007-9083-9. PMID 17533532
- [Background] Chan MR, Bedi S, Sanchez RJ, Young HN, Becker YT, Kellerman PS, Yevzlin AS. Stent placement versus angioplasty improves patency of arteriovenous grafts and blood flow of arteriovenous fistulae. Clin J Am Soc Nephrol. 2008 May;3(3):699-705. doi: 10.2215/CJN.04831107. Epub 2008 Feb 6. PMID 18256373
- [Background] Pan HB, Liang HL, Lin YH, Chung HM, Wu TH, Chen CY, Fang HC, Chen CK, Lai PH, Yang CF. Metallic stent placement for treating peripheral outflow lesions in native arteriovenous fistula hemodialysis patients after insufficient balloon dilatation. AJR Am J Roentgenol. 2005 Feb;184(2):403-9. doi: 10.2214/ajr.184.2.01840403. PMID 15671353
- [Background] Shemesh D, Goldin I, Zaghal I, Berlowitz D, Raveh D, Olsha O. Angioplasty with stent graft versus bare stent for recurrent cephalic arch stenosis in autogenous arteriovenous access for hemodialysis: a prospective randomized clinical trial. J Vasc Surg. 2008 Dec;48(6):1524-31, 1531.e1-2. doi: 10.1016/j.jvs.2008.07.071. Epub 2008 Oct 1. PMID 18829240
- [Background] Naoum JJ, Irwin C, Hunter GC. The use of covered nitinol stents to salvage dialysis grafts after multiple failures. Vasc Endovascular Surg. 2006 Aug-Sep;40(4):275-9. doi: 10.1177/1538574406291803. PMID 16959720
- [Background] Gupta M, Rajan DK, Tan KT, Sniderman KW, Simons ME. Use of expanded polytetrafluoroethylene-covered nitinol stents for the salvage of dysfunctional autogenous hemodialysis fistulas. J Vasc Interv Radiol. 2008 Jun;19(6):950-4. doi: 10.1016/j.jvir.2008.03.016. Epub 2008 Apr 28. PMID 18503914
- [Background] Clark TW, Rajan DK. Treating intractable venous stenosis: present and future therapy. Semin Dial. 2004 Jan-Feb;17(1):4-8. doi: 10.1111/j.1525-139x.2004.17103.x. PMID 14717801
- [Background] Yuan JG, Ohki T, Marin ML, Quintos RT, Krohn DL, Beitler JJ, Veith FJ. The effect of nonporous PTFE-covered stents on intimal hyperplasia following balloon arterial injury in minipigs. J Endovasc Surg. 1998 Nov;5(4):349-58. doi: 10.1583/1074-6218(1998)0052.0.CO;2. PMID 9867326
- [Background] Fontaine AB, Dos Passos S, Spigos D, Cearlock J, Urbaneja A. Use of polyetherurethane to improve the biocompatibility of vascular stents. J Endovasc Surg. 1995 Aug;2(3):255-65. doi: 10.1583/1074-6218(1995)0022.0.CO;2. PMID 9234140